CLINICAL TRIAL: NCT01076088
Title: A Phase III, Multicenter, Double-Blind, Randomized, Placebo-Controlled Clinical Trial in China to Study the Safety and Efficacy of Co-administration of Sitagliptin and Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Co-Administration of Sitagliptin and Metformin in China (MK-0431-121)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-121; 2010_514 (Other: Merck Registration Number)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sitagliptin 50 mg + metformin 500 mg (Experimental): Sitagliptin 50 mg and metformin 500 mg twice a day for 24 weeks.
  Interventions: Drug: Sitagliptin 50 mg; Drug: Metformin 500 mg
- Sitagliptin 50 mg + metformin 850 mg (Experimental): Sitagliptin 50 mg and metformin 850 mg twice a day for 24 weeks.
  Interventions: Drug: Sitagliptin 50 mg; Drug: Metformin 850 mg
- Metformin 500 mg (Active Comparator): Metformin 500 mg twice daily for 24 weeks.
  Interventions: Drug: Metformin 500 mg
- Metformin 850 mg (Active Comparator): Metformin 850 mg twice daily for 24 weeks.
  Interventions: Drug: Metformin 850 mg
- Sitagliptin 100 mg (Experimental): Sitagliptin 100 mg once daily for 24 weeks.
  Interventions: Drug: Sitagliptin 100 mg
- Placebo (Placebo Comparator): Matching placebo tablets for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin 50 mg — Sitagliptin 50 mg tablet twice a day, prior to the morning and evening meal, for 24 weeks.
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®
  Arms: Sitagliptin 50 mg + metformin 500 mg; Sitagliptin 50 mg + metformin 850 mg
Drug: Metformin 500 mg — Metformin 500 mg tablet twice daily, prior to the morning and evening meal, for 24 weeks.
  Other Names: Fortamet®, Glucophage®, Glucophage® XR, Glumetza®, Riomet®, Metgluco®, Glycoran®
  Arms: Metformin 500 mg; Sitagliptin 50 mg + metformin 500 mg
Drug: Sitagliptin 100 mg — Sitagliptin 100 mg once daily for 24 weeks.
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®
  Arms: Sitagliptin 100 mg
Drug: Placebo — Matching placebo tablets to sitagliptin or metformin for 24 weeks.
  Arms: Placebo
Drug: Metformin 850 mg — Metformin 850 mg tablet twice daily, prior to the morning and evening meal, for 24 weeks.
  Other Names: Fortamet®, Glucophage®, Glucophage® XR, Glumetza®, Riomet®, Metgluco®, Glycoran®
  Arms: Metformin 850 mg; Sitagliptin 50 mg + metformin 850 mg

SUMMARY:
This study will assess the efficacy and safety of initial treatment with sitagliptin and metformin in patients with type 2 diabetes mellitus in China. The primary hypothesis is that after 24 weeks, initial co-administration treatment with sitagliptin and metformin provided greater reduction in hemoglobin A1C (A1C) compared to initial treatment with sitagliptin alone and with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes mellitus
* is male, a female who cannot have children, or a female who agrees to use birth control during the study
* is not on an antihyperglycemic agent (AHA) (hemoglobin A1c [A1C] 7.5-11.0%) or on oral single AHA (A1C 7.0-10.5%) or low-dose AHA combination therapy (A1C 7.0-10.0%)

Exclusion Criteria:

* Patient has type 1 diabetes mellitus or ketoacidosis
* Patient is taking a dipeptidyl peptidase-4 (DPP-4) inhibitor (such as sitagliptin)
* Patient is on a weight loss program not in the maintenance phase or on a weight loss medication
* Patient has a history of liver disease, heart failure, heart disease, stroke, high blood pressure, blood disorders, or cancer
* Patient is HIV positive
* Patient is pregnant

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2012-12-24 (Actual); Study Completion 2012-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ji L, Han P, Wang X, Liu J, Zheng S, Jou YM, O'Neill EA, Golm GT, Engel SS, Kaufman KD, Shankar RR. Randomized clinical trial of the safety and efficacy of sitagliptin and metformin co-administered to Chinese patients with type 2 diabetes mellitus. J Diabetes Investig. 2016 Sep;7(5):727-36. doi: 10.1111/jdi.12511. Epub 2016 May 19. PMID 27181998

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 744 participants were randomized to treatment. Of these 744 participants, 1 participant, assigned to the placebo group, did not receive study medication. This participant was not included in the safety analyses.
Groups:
- Sitagliptin 50 mg + Metformin 500 mg: Sitagliptin 50 mg twice daily + metformin 500 mg twice daily
- Sitagliptin 50 mg + Metformin 850 mg: Sitagliptin 50 mg twice daily + metformin 850 mg twice daily
- Metformin 500 mg: Metformin 500 mg twice daily
- Metformin 850: Metformin 850 mg twice daily
- Sitagliptin 100 mg: Sitagliptin 100 mg once daily
- Placebo: Matching placebo to sitagliptin and/or metformin. Population includes 1 participant who did not receive any study medication.
Period: Overall Study
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 | Sitagliptin 100 mg | Placebo
Started | 122 | 125 | 126 | 124 | 120 | 127
Completed | 111 | 107 | 109 | 109 | 104 | 104
Not Completed | 11 | 18 | 17 | 15 | 16 | 23
Not completed — Adverse Event | 1 | 6 | 3 | 2 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 1 | 2
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 3 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 8 | 14 | 10 | 11 | 17
Not completed — Other protocol specified criteria | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 122 | 125 | 126 | 124 | 120 | 127 | 744
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (11.3) | 52.4 (9.3) | 52.6 (9.5) | 53.0 (10.3) | 51.7 (10.2) | 53.6 (9.7) | 52.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 58 | 57 | 49 | 46 | 40 | 287
  Male | 85 | 67 | 69 | 75 | 74 | 87 | 457
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin] | 8.46 (0.97) | 8.66 (0.95) | 8.69 (0.99) | 8.67 (1.08) | 8.74 (1.14) | 8.97 (1.05) | 8.70 (1.04)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 175.6 (40.6) | 181.9 (43.0) | 184.6 (46.8) | 183.5 (47.7) | 182.5 (44.0) | 185.8 (47.3) | 182.3 (45.0)
2-hour post meal glucose (2-h PMG) [Mean (Standard Deviation); unit: mg/dL] — Participants with data: sita50/met500, n=121; sita50/met850, n=125; met500, n=125; met850, n=123; sita100, n=119; placebo; n=126; total, n=739
  mg/dL | 292.7 (81.2) | 292.9 (68.4) | 303.2 (74.1) | 298.8 (74.6) | 297.7 (74.7) | 308.3 (83.6) | 299.0 (76.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 24
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 24
Population: Full Analysis Set, all randomized participants except those who: failed to take at least 1 dose of study treatment, lacked all post-randomization data for the A1C subsequent to at least 1 dose of study treatment, or lacked baseline data for the A1C. Last observation carried forward (missing data approach).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin
Groups:
- Metformin 850 mg: Metformin 850 mg twice daily
- Placebo: Matching placebo to sitagliptin and/or metformin
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 118 | 114 | 116 | 117 | 113 | 117
Percent of glycosylated hemoglobin | -1.67 [-1.92 to -1.43] | -1.83 [-2.07 to -1.58] | -1.29 [-1.54 to -1.04] | -1.56 [-1.80 to -1.32] | -0.99 [-1.24 to -0.75] | -0.59 [-0.84 to -0.34]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Metformin 850 mg; Test type: Superiority or Other; p = 0.087, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. metformin 850 mg. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior antihyperglycemic agent (AHA) therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.27, 95% CI 2-sided [-0.58 to 0.04]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. sitagliptin 100 mg. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.84, 95% CI 2-sided [-1.15 to -0.52]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Metformin 500 mg; Test type: Superiority or Other; p = 0.014, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. metformin 500 mg. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.39, 95% CI 2-sided [-0.69 to -0.08]
Statistical Analysis 4: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. sitagliptin 100 mg. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.68, 95% CI 2-sided [-0.99 to -0.37]
Statistical Analysis 5: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. placebo. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -1.24, 95% CI 2-sided [-1.55 to -0.93]
Statistical Analysis 6: Comparison: Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 850 mg vs. placebo. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.97, 95% CI 2-sided [-1.28 to -0.66]
Statistical Analysis 7: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. placebo. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -1.08, 95% CI 2-sided [-1.39 to -0.78]
Statistical Analysis 8: Comparison: Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 500 mg vs. placebo. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.70, 95% CI 2-sided [-1.01 to -0.39]
Statistical Analysis 9: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — Pairwise comparison, sitagliptin 100 mg vs. placebo. The normality assumption required for validity of ANCOVA was violated due to a biologically implausible extreme outlier. See below for results using robust regression; The ANCOVA model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in Least Squares Mean = -0.40, 95% CI 2-sided [-0.71 to -0.09]
Statistical Analysis 10: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Metformin 850 mg; Test type: Superiority or Other; p = 0.008, Regression, Robust — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. metformin 850 mg. This is a post-hoc analysis using robust regression, a valid method in the presence of outliers; The Robust Regression model included terms for treatment and prior AHA therapy status (yes/no) and a covariate for baseline A1C; Difference in least squares mean = -0.36, 95% CI 2-sided [-0.62 to -0.09]
Statistical Analysis 11: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Robust — Comparing co-administration with individual components. This is a post-hoc analysis using robust regression, a valid method in the presence of outliers; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.87, 95% CI 2-sided [-1.13 to -0.60]
Statistical Analysis 12: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Metformin 500 mg; Test type: Superiority or Other; p = 0.007, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.36, 95% CI 2-sided [-0.63 to -0.10]
Statistical Analysis 13: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.61, 95% CI 2-sided [-0.88 to -0.35]
Statistical Analysis 14: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -1.25, 95% CI 2-sided [-1.52 to -0.99]
Statistical Analysis 15: Comparison: Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.90, 95% CI 2-sided [-1.16 to -0.63]
Statistical Analysis 16: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -1.00, 95% CI 2-sided [-1.26 to -0.74]
Statistical Analysis 17: Comparison: Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.64, 95% CI 2-sided [-0.90 to -0.37]
Statistical Analysis 18: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Robust — [p-value comment as in outcome 1, analysis 11]; [statistical method as in outcome 1, analysis 10]; Difference in Least Squares Mean = -0.39, 95% CI 2-sided [-0.65 to -0.12]

2. Secondary Outcome: Change From Baseline in 2-hour Post Meal Glucose (2-h PMG) at Week 24
Description: Change from baseline in 2-h PMG at Week 24 is defined as Week 24 2-h PMG minus Week 0 2-h PMG.
Time Frame: Baseline and Week 24
Population: Full Analysis Set, all randomized participants except those who: failed to take at least 1 dose of study treatment, lacked all post-randomization data for 2-h PMG subsequent to at least 1 dose of study treatment, or lacked baseline data for 2-h PMG. Last observation carried forward (missing data approach).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 110 | 110 | 112 | 108 | 107 | 107
mg/dL | -97.05 [-109.01 to -85.09] | -109.46 [-121.47 to -97.44] | -65.67 [-77.76 to -53.58] | -90.93 [-103.04 to -78.83] | -48.11 [-60.37 to -35.85] | -21.88 [-34.33 to -9.43]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Metformin 850; Test type: Superiority or Other; p = 0.017, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. metformin 850 mg; The ANCOVA model included terms for treatment and prior antihyperglycemic agent (AHA) therapy status (yes/no) and a covariate for baseline 2-H PMG; Difference in Least Squares Mean = -18.52, 95% CI 2-sided [-33.75 to -3.29]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. sitagliptin 100 mg; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -61.34, 95% CI 2-sided [-76.61 to -46.07]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Metformin 500 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. metformin 500 mg; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -31.38, 95% CI 2-sided [-46.49 to -16.28]
Statistical Analysis 4: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. sitagliptin 100 mg; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -48.94, 95% CI 2-sided [-64.21 to -33.67]
Statistical Analysis 5: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. placebo; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -87.57, 95% CI 2-sided [-102.87 to -72.27]
Statistical Analysis 6: Comparison: Metformin 850 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 850 mg vs. placebo; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -69.05, 95% CI 2-sided [-84.41 to -53.70]
Statistical Analysis 7: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. placebo; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -75.17, 95% CI 2-sided [-90.47 to -59.87]
Statistical Analysis 8: Comparison: Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 500 mg vs. placebo; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -43.79, 95% CI 2-sided [-58.99 to -28.58]
Statistical Analysis 9: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 100 mg vs. placebo; [statistical method as in outcome 2, analysis 1]; Difference in Least Squares Mean = -26.23, 95% CI 2-sided [-41.62 to -10.84]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline in FPG at Week 24 is defined as Week 24 FPG minus Week 0 FPG.
Time Frame: Baseline and Week 24
Population: Full Analysis Set, all randomized participants except those who: failed to take at least 1 dose of study treatment, lacked all post-randomization data for FPG subsequent to at least 1 dose of study treatment, or lacked baseline data for FPG. Last observation carried forward (missing data approach).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 118 | 116 | 119 | 119 | 114 | 119
mg/dL | -39.38 [-46.29 to -32.47] | -47.74 [-54.73 to -40.75] | -33.66 [-40.66 to -26.66] | -39.63 [-46.50 to -32.76] | -21.86 [-28.92 to -14.80] | -11.93 [-18.94 to -4.92]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Metformin 850; Test type: Superiority or Other; p = 0.069, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. metformin 850 mg; The ANCOVA model included terms for treatment and prior antihyperglycemic agent (AHA) therapy status (yes/no) and a covariate for baseline FPG; Difference in Least Squares Mean = -8.11, 95% CI 2-sided [-16.86 to 0.64]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. sitagliptin 100 mg; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -25.88, 95% CI 2-sided [-34.72 to -17.04]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Metformin 500 mg; Test type: Superiority or Other; p = 0.198, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. metformin 500 mg; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -5.72, 95% CI 2-sided [-14.44 to 3.00]
Statistical Analysis 4: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. sitagliptin 100 mg; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -17.53, 95% CI 2-sided [-26.33 to -8.72]
Statistical Analysis 5: Comparison: Sitagliptin 50 mg + Metformin 850 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 850 mg vs. placebo; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -35.81, 95% CI 2-sided [-44.56 to -27.06]
Statistical Analysis 6: Comparison: Metformin 850 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 850 mg vs. placebo; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -27.70, 95% CI 2-sided [-36.40 to -19.00]
Statistical Analysis 7: Comparison: Sitagliptin 50 mg + Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, sitagliptin 50 mg + metformin 500 mg vs. placebo; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -27.45, 95% CI 2-sided [-36.18 to -18.73]
Statistical Analysis 8: Comparison: Metformin 500 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison, metformin 500 mg vs. placebo; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -21.73, 95% CI 2-sided [-30.42 to -13.04]
Statistical Analysis 9: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.027, ANCOVA — Pairwise comparison, sitagliptin 100 mg vs. placebo; [statistical method as in outcome 3, analysis 1]; Difference in Least Squares Mean = -9.93, 95% CI 2-sided [-18.72 to -1.14]

ADVERSE EVENTS:
Description: All participants as treated population. Serious and non-serious adverse events (AEs) include and exclude data after rescue therapy, respectively. One event of hypoglycaemia that, per protocol, should have been reported as an AE was not reported as an AE. This event occurred in a participant who had another event of hypoglycaemia that was reported.
Groups:
- Placebo: Matching placebo to sitagliptin and/or metformin. Population excludes 1 participant who did not receive any study medication.
Arm/Group | Sitagliptin 50 mg + Metformin 500 mg | Sitagliptin 50 mg + Metformin 850 mg | Metformin 500 mg | Metformin 850 | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/125 | 1/126 | 1/124 | 3/120 | 1/126
Other Adverse Events (participants affected / at risk) | 9/122 | 14/125 | 8/126 | 13/124 | 6/120 | 4/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 50 mg + Metformin 500 mg (N=122) | Sitagliptin 50 mg + Metformin 850 mg (N=125) | Metformin 500 mg (N=126) | Metformin 850 (N=124) | Sitagliptin 100 mg (N=120) | Placebo (N=126)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulation time shortened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 50 mg + Metformin 500 mg (N=122) | Sitagliptin 50 mg + Metformin 850 mg (N=125) | Metformin 500 mg (N=126) | Metformin 850 (N=124) | Sitagliptin 100 mg (N=120) | Placebo (N=126)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 4 (4) | 9 (10) | 2 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (10) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 7 (11) | 3 (3) | 2 (2) | 4 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.